CLINICAL TRIAL: NCT05842356
Title: Parental Feelings About Their Child Needing a Central Line
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jeffrey D. Edwards, Associate Professor of Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AAAU3577
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Critical Illness; Children, Only; Stress
Keywords: Central Venous Line (CVL); Peripherally Inserted Central Catheter (PICC)
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants (parents) will not know which communication technique group they are in until after their participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication Technique 1 (No Intervention): A standard communication technique will be used in this group.
- Communication Technique 2 (Experimental): A new communication technique will be used in this group.
  Interventions: Behavioral: Communication Technique 2

INTERVENTIONS:
Behavioral: Communication Technique 2 — A new communication technique.
  Arms: Communication Technique 2

SUMMARY:
The goal of this research project is to determine if different communication techniques during the consent process impact parental anxiety and comfort providing consent.

DETAILED DESCRIPTION:
The parents of children in the pediatric intensive care units (PICUs) at Columbia University may be asked if they are interested in participating in this study if their child needs a central venous line (CVL) or peripherally inserted central catheter (PICC) placed.

If the parents are interested in participating, they will be randomly assigned to a communication technique group while they are discussing the procedure and giving consent with a medical team member. After they provide consent, they will be asked to complete surveys about their thoughts and feelings. The study should take about 15 minutes.

After data is collected, the researchers will compare survey answers between the two communication styles used with parents.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian of a child admitted to the pediatric intensive care units (PICUs) at Columbia University
* The child needs a central venous line (CVL) or peripherally inserted central catheter (PICC) placed in the PICU
* The parent or guardian speaks English or Spanish

Exclusion Criteria:

* Parents or guardians who speak languages other than English or Spanish
* Parents or guardians of children who need a CVL or PICC placed during an emergency without consent
* Parents or guardians who are unable to be physically present and provide consent over the phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-13 (Actual)

PRIMARY OUTCOMES:
Parental Anxiety | 15 minutes
  The parental anxiety survey is a tool used to measure levels of parental anxiety at the time of consent. Scores range from 7 to 28 with lower scores representing lower levels of anxiety.
Parental Comfort Providing Consent | 15 minutes
  The parental comfort providing consent survey score is a tool used to measure parental comfort in providing consent. Scores range from 0 to 24 with lower scores representing higher levels of comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Edwards, MD, MA, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University New York-Presbyterian Morgan Stanley Children's Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No